CLINICAL TRIAL: NCT07065344
Title: A Multicenter Observational Study to Understand the Clinical Characteristics, Treatment Patterns and Access to Novel Therapies of Patients With Diffuse Large B-Cell Lymphoma in the MEA Region A Cross-sectional Multi-center, Observational Study to Describe the Disease Characteristics and Treatment Patterns and Explore Access to Novel Therapies for Diffuse Large B-Cell Lymphoma (DLBCL) Patients for Both Treatment naïve and Relapsed/Refractory Patients in the Middle East & Africa (MEA) Region.
Brief Title: A Multicenter Observational Study to Understand the Clinical Characteristics, Treatment Patterns and Access to Novel Therapies of Patients With Diffuse Large B-Cell Lymphoma in the MEA Region
Acronym: DOMAIN
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00080
Record Dates: First submitted 2025-05-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hematology; Diffused Large B Cell Lymphoma
Keywords: Diffused Large B Cell Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- - Cohort 1: Treatment naïve, treatment-eligible (according to investigator's decision) DLBCL.: 333 patients treatment naïve, treatment-eligible DLBCL patients
- - Cohort 2: Relapsed/Refractory DLBCL who have failed at least one prior therapy.: 167 patients relapsed and/or refractory DLBCL patients who have failed at least one prior therapy.

SUMMARY:
Non-Hodgkin lymphoma (NHL) is the most common hematologic malignancy, with over 80,500 estimated new cases diagnosed in the United States in 20231. Diffuse large B-cell lymphoma (DLBCL) is the most frequent subtype of NHL, accounting for 30%-40% of cases2. DLBCL is an aggressive malignancy with heterogeneous biology and behavior. Disease risk stratification and treatment planning involve various patient and clinical characteristics (e.g., age, stage, and tumor bulk), prognostic indices (e.g., International Prognostic Index (IPI) score), and gene expression profiling. Patients typically present with nodal or extranodal disease, usually exhibiting rapid tumor growth and symptoms that are highly dependent upon the tumor localization.

The diagnosis and subtyping of DLBCL have significantly advanced, from morphological assessment of tissue slide to numerous ancillary tests, including immunophenotyping performed by immunohistochemistry (IHC), cytogenetics, and detailed molecular testing to classify the disease based on cell of origin (COO). With the advent of novel therapeutic options, molecular subtyping of DLBCL at diagnosis is expected to allow prognostic stratification of patients into distinct subgroups. This stratification could provide a preclinical rationale for therapeutic targeting the involved pathways and paving the application of personalized treatment.

DLBCL is a potentially curable disease with an overall 60-70% chance of achieving durable complete remission (CR) with the currently used standard first-line immunochemotherapy. However, 30-40% of patients are either refractory to first-line treatment or experience relapse and eventually will die of disease progression7. Although high-dose chemotherapy followed by autologous stem cell transplant (ASCT) is the recommended SOC for eligible patients in the second-line setting based on results from the pivotal PARMA study, real-world SOC in this setting remains less clearly defined.

Patients not cured with ASCT or ineligible to ASCT or refractory to salvage chemotherapy may be considered for Chimeric Antigen Receptor (CAR) T cell therapy targeting CD1910. Although ASCT and CAR-T cell therapy offer patients an opportunity for durable remission, many patients may not be eligible for ASCT or CAR-T cell therapy or relapse after these treatments. In the last decade, the investigation of novel antigens, which can be targeted by immunotherapy and identified to eliminate malignant cells regardless of their molecular pathogenesis, has been constantly pursued.

This study aims to address this need by examining the demographic, clinical characteristics, and treatment patterns and exploring access to novel therapies for diffuse large B-cell lymphoma (DLBCL) patients, both treatment naïve and relapsed/refractory patients, in the Middle East and Africa (MEA) region.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older at diagnosis.
2. Patients who have confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) according to the investigator's decision and/or histopathological diagnosis.
3. For Cohort 1: DLBCL patients who are eligible to start treatment* according to the investigator's decision.
4. For Cohort 2: patients who are diagnosed with DLBCL and have failed at least one prior line of therapy.
5. Patients willing to sign the written informed consent form (ICF) indicating that they understand the purpose of the study and procedures required for participation.

Exclusion Criteria:

1. Patients who are not eligible for treatment for any reason, according to the investigator's judgment and decision
2. Patients with concurrent active malignancies other than DLBCL.
3. Patients who are actively participating in any other clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to recruit approximately 500 patients, divided as follows:
  * Cohort 1: 333 patients treatment naïve, treatment-eligible DLBCL patients.
  * Cohort 2: 167 patients relapsed and/or refractory DLBCL patients who have failed at least one prior therapy.
  Patients will be selected based on strict inclusion and exclusion criteria to ensure the validity and reliability of the study results. The study will be conducted across eight countries in the Middle East and Africa (MEA) region, including Egypt, South Africa, Turkey, Iraq, Morocco, and the Gulf Cooperative Council (GCC), including the Kingdom of Saudi Arabia (KSA), the United Arab Emirates (UAE), and Kuwait.
  Approximately 15-20 sites within these countries will participate in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To describe the treatment patterns for the first line and subsequent therapies for DLBCL patients | 22 months
  ▪ Type of regimen: Chemoimmunotherapy "CIT" and regimen name, targeted therapies and name, bone marrow transplantations (BMT), T-cell engagers and name, and CAR-T cell therapy and name, Antibody Drug Conjugate (ADC) and Name, Anti-CD79b (Polatuzumab), Anti-CD-19 (Tafasitamab).

SECONDARY OUTCOMES:
To describe the patient demographics and disease characteristics of DLBCL patients | 22 Months
  - Patient demographics:
  * Age
  * Gender
  * Ethnicity
To identify and characterize patients according to risk profiles | 22 Months
  Describing patients' risk profiles, including:
  - Cytogenetic aberrations
To explore access to novel therapies for DLBC | 22 Months
  Exploring access to novel therapies for DLBCL:
  ▪ Proportion (%) of patients receiving the prescribed novel therapies
Describing patients' risk profiles | 22 Months
  Immunohistochemistry results (Positive/Negative/Unknown)